CLINICAL TRIAL: NCT04276701
Title: Immune Mediators and Metabolites to Stratify Systemic Lupus Erythematosus Patients at High Risk of Cardio Vascular Diseases
Acronym: ISLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Foundation for Research in Rheumatology (FOREUM) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2019/38
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Immune mediators; Immune metabolites; cardio vascular diseases; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic lupus erythematosus (SLE) (Experimental)
  Interventions: Biological: blood sample; Other: Ultrasonography assessment; Behavioral: questionnaires

INTERVENTIONS:
Biological: blood sample — 35 ml whole blood for Peripheral blood mononuclear cell (PBMC), serum and plasma
Other: Ultrasonography assessment — assessment of atherosclerotic plaques and measurement of carotid intima-media thickness (cIMT)
Behavioral: questionnaires — Food and exercise questionnaires validated by the American heart Association

SUMMARY:
Accelerated atherosclerosis is an established complication of systemic autoimmune diseases, particularly SLE. Young female patients with SLE are more likely to develop myocardial infarction than matched healthy controls, and CVD is nowadays one of the most common causes of death (27%) in lupus patients. While traditional CV risk factors cannot explain such increased CV morbidity associated with SLE, common disease factors shared between SLE, atherosclerosis and treatment exposure may be of outmost importance in this process. Our group made 3 findings of particular interest that could link SLE pathogenesis and atherosclerosis-associated immune dysregulation: 1/ the investigators identified specific immunometabolites (circulating nucleotide-derived metabolites adenine and N4-acetylcytidine), which are increased in the circulation of SLE patients. These immunometabolites trigger a constitutive inflammasome activation resulting in aberrant IL1-β production. Given that IL1-β inhibition was reported to significantly reduce CV events without altering lipid levels, the investigators propose that these immunometabolites may represent novel candidate biomarkers of CV risk stratification in SLE. 2/ the investigators identified OX40L as an important costimulatory molecule implicated in follicular helper T cell (Tfh) activation in SLE. Interestingly, OX40L polymorphism has been associated to both SLE and atherosclerosis, and Tfh have been recently shown to accelerate atherosclerosis progression. 3/ Immune complexes-activated platelets sustain aberrant immune response in SLE and block immunosuppressive functions of regulatory T cells (Tregs) in a P-selectin/PSGL1 dependent manner. Selectins and Tregs cell dysfunction are well accepted players in atherosclerosis pathogenesis.

Thus there are multiple pathways that are shared between SLE and atherosclerosis and that may results in an increased risk of CV-associated morbidity in SLE patients. Exploring these interconnected pathways in SLE patients together with traditional and other well-established disease-related factors, might lead to a better stratification of CV risk in SLE.

The aim of this study is to investigate the accuracy, predictive value and utility of immunological disease-related biomarkers in stratifying CV risk in patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged over 18 years old.
* SLE diagnosis according to the 2019 European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) Classification Criteria for Systemic Lupus Erythematosus
* Having signed an informed consent (at the latest on the day of inclusion and before any examination required by research).

Exclusion Criteria:

* Pregnancy or breast-feeding for woman.
* Person concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who show atherosclerotic plaque progression defined by the absence of carotid plaque in patients at baseline and its subsequent development at follow-up evaluated by semi-automated 3D vascular ultrasound | At baseline (Day 0) and 18 months from baseline

SECONDARY OUTCOMES:
Proportion of patients who show carotid Intima Media Thickness (cIMT) progression measured in the common carotid artery, at the bulb and the origin of the internal carotid artery | At baseline (Day 0) and 18 months from baseline
  defined as an increase of 0.1mm or more evaluated by vascular ultrasound.
Proportion of patients with atherosclerotic plaques | At baseline (Day 0) and 18 months from baseline
Proportion of patients with hypertension | At baseline (Day 0) and 18 months from baseline
Proportion of patients with Body Mass Index around 30 or more | At baseline (Day 0) and 18 months from baseline
Proportion of patients who are smokers or past-smokers | At baseline (Day 0) and 18 months from baseline
Proportion of patients who present a history of ischemic heart disease | At baseline (Day 0) and 18 months from baseline
Proportion of patients who present a history of cerebral vascular accident | At baseline (Day 0) and 18 months from baseline
Proportion of patients who present a history of peripheral artery disease | At baseline (Day 0) and 18 months from baseline
Change in waist size in centimeters | At baseline (Day 0) and 18 months from baseline
Change in blood glucose levels in milligram per deciliter | At baseline (Day 0) and 18 months from baseline
Change in total cholesterol levels | At baseline (Day 0) and 18 months from baseline
Change in HDL cholesterol levels | At baseline (Day 0) and 18 months from baseline
Change in LDL cholesterol levels | At baseline (Day 0) and 18 months from baseline
Change in triglycerides levels | At baseline (Day 0) and 18 months from baseline
Change in Very Low Density Lipoprotein (VLDL) levels | At baseline (Day 0) and 18 months from baseline
Change in C-Reactive protein levels | At baseline (Day 0) and 18 months from baseline
Change in insulin levels | At baseline (Day 0) and 18 months from baseline
Change in lupus disease activity according to Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | At baseline (Day 0) and 18 months from baseline
  score (Min value: 0 - Max value: 105), with higher values mean higher disease activity.
Change in lupus disease activity according to Systemic Lupus International Collaborating Clinics /American College of Rheumatology (SLICC/ACR) damage index | At baseline (Day 0) and 18 months from baseline
  (Min value: 0 - Max value: 47), with higher values mean more important damages.
Change in glucocorticoids intake | At baseline (Day 0) and 18 months from baseline
Change in platelets-derived biomarkers (P-selectin, sCD154) in micrograms per milliliter, evaluated by Western Blot analysis. | At baseline (Day 0) and 18 months from baseline
Change in neutrophils-derived biomarkers Proteins S100A8, A9, A8/9, and A12, IL-6 in micrograms per milliliter, evaluated by Western Blot analysis. | At baseline (Day 0) and 18 months from baseline
Change in interleukin-6 levels | At baseline (Day 0) and 18 months from baseline
Change in interleukin-12 levels | At baseline (Day 0) and 18 months from baseline
Change in T-Follicular Helpers lymphocytes | At baseline (Day 0) and 18 months from baseline
Change in myeloperoxidase-conjugated DNA levels in fluorescence intensity evaluated by fluorometric assay. | At baseline (Day 0) and 18 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DUFFAU, Prof, Principal Investigator — University Hospital, Bordeaux; Patrick BLANCO, Prof, Study Director — University Hospital, Bordeaux
Locations (6):
- France (5):
  - CHU de Bordeaux - service de médecine interne, Bordeaux
  - CHU de Brest - service de rhumatologie, Brest
  - CHRU de Lille - service de Médecine Interne, Lille
  - AP-HP - Hôpital Cochin - service de Médecine Interne, Paris
  - CHU de Strasbourg - service d'Immunologie Clinique, Strasbourg
- Universität Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No